CLINICAL TRIAL: NCT04643366
Title: Phase 2 Study of Total Neoadjuvant mFOLFOX and Short-Course Radiotherapy in Resectable Rectal Cancer
Brief Title: Total Neoadjuvant Therapy With mFOLFOX and Short-course Radiation in Resectable Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18-14260; HM20020384 (Other: Virginia Commonwealth University); NCI-2020-13796 (Other: NCI CTRP)
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: Resectable; Rectal
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Concurrent Chemotherapy/ Radiation Therapy (Experimental): 5-Fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6) four 14-day cycles will be given before CRT starts. Pelvic Intensity-modulated radiation therapy (IMRT): 25 Gy in 5 fractions over 5 days + Continuous infusion 5-fluorouracil (5-FU) for 4 days (96 hours) followed by four 14-day cycles of (mFOLFOX6) to be given after CRT ends.
  Interventions: Drug: Chemotherapy; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Chemotherapy — Neoadjuvant chemotherapy with 2 months of combination oxaliplatin and 5-Fluorouracil, leucovorin, and oxaliplatin (mFOLFOX)
Radiation: Radiation Therapy — Pelvic Intensity-modulated radiation therapy (IMRT)

SUMMARY:
This is phase 2 trial of neoadjuvant therapy and short-course radiotherapy in resectable rectal cancer.

DETAILED DESCRIPTION:
This trial involves 4 cycles of systemic chemotherapy followed by short-course RT with concurrent 5-FU neoadjuvant chemoradiotherapy (CRT) and subsequent consolidation with 4 cycles of systemic chemotherapy prior to surgery or, for those who achieve cCR, the option of non-operative active surveillance.Three-year disease free survival (DFS) defined as the percentage of patients alive without recurrence of disease at 3 years measured from the date of clinical complete response (cCR) or date of total mesorectal excision (TME) at surgery (whichever is earlier).

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of adenocarcinoma of the rectum (diagnosis by tissue biopsy) within 90 days prior to registration. At least a portion of the tumor must be located below the peritoneal reflection or begin within 12 cm of the anal verge on flexible endoscopy
* Clinically staged (AJCC 8th ed.) T3-4 N0 M0 or T any N1-2 M0 based upon the following minimum diagnostic workup:

  * Colonoscopy, unless patient presents with an obstructing lesion
  * Within 30 days prior to registration:
* History/physical examination
* Imaging to exclude distant metastases: either contrast-enhanced CT of the chest, abdomen, and pelvis or whole-body PET-CT or MRI
* Pelvic MRI (preferred) or transrectal ultrasound (TRUS) for T staging Note: Patients may have initiated standard mFOLFOX6 treatment before study registration provided that they met the above criteria before initiating treatment and can feasibly continue to CRT according to the timeline described in Section
* ECOG Performance Status ≤2
* Age ≥ 18 years
* Adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,200 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥8.0 g/dL is acceptable.)
* Adequate liver and renal function defined as follows:

  * AST and alkaline phosphatase < 2.5 x upper limit of normal (ULN)
  * Bilirubin ≤ 2.5 ULN
  * Calculated creatinine clearance (CrCl) > 30 mL/min using Cockcroft-Gault formula as calculated by the standard Cockcroft-Gault equation using age, actual weight, creatinine, and gender
* Must be deemed a candidate for curative resection by the surgical oncologist who will be performing the operation
* Women of childbearing potential (WCBP) must have a negative serum pregnancy test performed within 7 days prior to the start of chemotherapy.
* WCBP and men must agree to use a medically accepted form of birth control during the treatment and for 3 months following completion of chemotherapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior RT that would result in unsafe overlap of RT fields with the planned study treatment, per the treating radiation oncologist
* Clinically significant cardiac disease, including major cardiac dysfunction, that in the opinion of the treating medical oncologist would preclude them from receiving systemic therapy with 5-fluorouracil, leucovorin or oxaliplatin.
* Serious (ie, ≥ grade 3) uncontrolled infection
* Pulmonary or respiratory condition that, in the opinion of the treating medical oncologist would preclude them from receiving systemic therapy with 5-fluorouracil, leucovorin or oxaliplatin.
* Major surgery within 28 days of study enrollment (other than diverting colostomy)
* History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis) requiring significant intervention (eg, hospitalization, surgery, immunosuppressive medications) that would, in the opinion of the investigator, preclude study therapy
* Prior known allergic reaction to 5-fluorouracil, leucovorin, or oxaliplatin
* Known dipyrimidine dehydrogenase deficiency (DPD)
* Any evidence of distant metastases (M1)
* Pregnant or breast feeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Three-year disease free survival (DFS) | 3 years after end of treatment
  The three-year disease free survival (DFS) defined as the number of patients alive without recurrence of disease at 3 years measured from the date of clinical complete response (cCR) or date of total mesorectal excision (TME) at surgery (whichever is earlier).

SECONDARY OUTCOMES:
Pathologic complete response (pCR) rate | 3 Years after end of treatment
  The number of patients that achieve pathologic complete response(pCR)(defined as negative surgical margins and no evidence of residual viable tumor) at time of total mesorectal excision (TME).
Clinical complete response (cCR) following total neoadjuvant therapy (TNT) based on tumor response | 3 Years after end of treatment
  Determine the cCR using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), in patients evaluable for response
The number of Adverse events (AEs) per participant | 39 Months
  The number of Adverse events (AEs) per participant characterized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v. 5.0)
Progression (PFS) Rate | 3 Years after end of treatment
  PFS defined as the time from initiation of chemotherapy until date of progression
Overall Survival (OS) Rate | 3 Years after end of treatment
  OS defined as the time from initiation of chemotherapy until death by any cause.
Number of patients who do not require an ostomy at time of surgery | 116 Days
  After neoadjuvant therapy is complete patients will undergo assessment of disease status prior to determination of whether they will proceed to surgical resection or active surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Matin, MD, Principal Investigator — Massey Cancer Center
Locations (3):
- United States (3):
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Healthcenter, South Hill, Virginia

IPD SHARING:
Plan to Share IPD: No